CLINICAL TRIAL: NCT03117088
Title: Safe-SCOPE Pilot Study: Standardized Checklist Of Patient Information Exchange
Brief Title: Safe-SCOPE Pilot Study
Acronym: Safe-SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CTCA-16-164
Record Dates: First submitted 2017-03-14; First posted 2017-04-17 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Quality Assurance of Patient Safety
Keywords: Standardized handover; Online-based; SOFA-Score; ICU; ISBAR3

STUDY DESIGN:
Intervention Model Description: two armed cluster randomized crossover three periods prospective single centre pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Checklist ISBAR 3 (Active Comparator): online-based checklist for standardized handovers
  Interventions: Other: Checklist ISBAR3
- Checklist VICUR (Placebo Comparator): comparator Checklist
  Interventions: Other: Checklist VICUR

INTERVENTIONS:
Other: Checklist ISBAR3 — Checklist ISBAR 3
  Use of an online based checklist for handovers with the following items:
  Identification Situation Background Assessment Recommendation Read- back Risk
  Established Checklist as communication tool
  Arms: Checklist ISBAR 3
Other: Checklist VICUR — Checklist Vicur
  Use of an online based alternative checklist for handovers with the following items:
  Vaccination status Insurance status Contact person Utilisation Rehabilitation Organ donor? Patient decree?
  alternative checklist missing communication tool
  Arms: Checklist VICUR

SUMMARY:
Study Title Safe- SCOPE Pilot Study Standardized Checklist of Patient Information Exchange

Short Title Safe- SCOPE Pilot Study

Study Design: Single centre two armed cluster randomised crossover pilot study

Study duration: 5 months

Objectives:

* Influence of standardised checklists on medical/ physician handovers on an Intensive Care Unit -ICU and its influence on patient safety
* Satisfaction survey in physicians group

Number of patients:

All patients treated on OIM during assessment period

Checklist Intervention

* All physicians working in the department of Intensive Care Medicine and Intermediate Care are informed and enlightened about Safe-SCOPE Pilot Study. After written consent participating physicians will use an online form ISBAR3 Checklist or alternative Checklist for handovers twice a day.
* Handover times/schedule:

OIM 1,2,3,5, und 6: 7:30 am and 7:30 pm OIM 4 und WEA 1: 7:30 am and 2:00 pm

* ISBAR3 Checklist
* VICUR Checklist wash- out Phase:
* No checklists for one month

Efficacy:

Patients:

* Mortality rate
* Duration on ICU
* Reuptake on ICU
* SOFA Score on admission to ICU, 48h, 72h and 120h after admission
* Handover duration per patient
* Number of enclosed patients

Handover:

* Entire handover duration
* Interruptions during handover

DETAILED DESCRIPTION:
The simplest definition of patient safety is the prevention of errors and adverse events to patient associated with health care. While health care has become more effective it has also become more complex, with greater use of new technologies, medicines and treatments. Health services treat older and sicker patients who often present with significant co- morbidities requiring more and more difficult decisions as to health care priorities.

European data, mostly from European Union Member States, consistently show that medical errors and health care related adverse events occur in 8-12% of hospitalization. For example, the United Kingdom Department of health, in its 2000 report "An organisation with a memory", estimated about 850 000 adverse events a year (10% of hospital admissions). Spain (in its 2005 national study of adverse events) and France and Denmark have published incidence studies with similar results.

While 23% of European Union citizens claim to have been directly affected by medial errors, 18% claim to have experienced a serious medical error in a hospital and 11% to be prescribed wrong medication. Evidence on medial errors shows that 50% to 70,2% of such harm can be prevented through comprehensive systematic approaches to patient safety.

Statistics of the World Health Organisation (WHO) show further more that strategies to reduce the rate of adverse events in the European Union alone would lead to the prevention of more than 750 000 harm-inflicted medial errors per year, leading in turn to over 3,2 million fewer days of hospitalization, 260 000 fewer incidents of permanent disability, and 95 000 fewer deaths per years. Our working group clarifies this as very impressive data and statistics.

In aviation checklists are an established instrument to avoid adverse events and so to improve safety. Like in the cockpit also in operating room checklists and briefings can be useful to reduce perceived risks and improve collaboration among operating rooms personnel by controlling safety standards, availability of required sources and responsibility assignment. The World Health Organisation WHO in 2009 established checklist (Save Surgery Saves Lives) is a feasible task increasingly used with individual adaptation. The Implementation has to be ingrained in a hospital wide safety culture with patient safety- related behaviour and perceived personal empowerment. The safe surgery saves lives campaign showed in eight hospitals worldwide with different socio- ecological backgrounds that in around 8. 000 operations mortality and infections rate decreased significantly after using the safe surgery saves lives checklist in operating theatres.

Checklists are efficient working tools used as a reminder or to structure processes. They guarantee that processes are objective and reproducible and therefore increase patient- safety. Especially in stress and emergency situations as they exist on an Intensive Care Unit checklists can help to avoid mind mistakes and demonstrate possible decisions.

Related to these data and statistics and on that important background we are planning a multi-centre main trial on improving patient safety: Standardized Checklist of Patient Information Exchange. Because there is no information about the magnitude of checklist effects on patient data and there is no risk for the patients we use the Safe SCOPE Pilot study to estimate the effects size of the checklists and to investigate the feasibility of the main trial.

ELIGIBILITY:
Inclusion Criteria:

Physicians:

* all physicians working on ICU (department of Intensive Medicine and Intermediate Care) during data collection
* existing written consent

Patients:

* All patients treated in the department of Intensive Care Medicine and Intermediate Care (OIM) during assessment period who passed at least two online form based handovers

Exclusion Criteria:

Physicians:

* missing written consent
* Chief of the department of Intensive Care medicine and Intermediate Care
* Colleagues involved in Safe- SCOPE Pilot Study protocol or group of experts

Patients:

* Age < 18 years
* Pregnancy
* ward shift within OIM and hereby associated cluster change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change of SOFA Score at hour 48 | admission and hour 48
  Change of SOFA Score to baseline (admission) and 48 hours after admission

SECONDARY OUTCOMES:
Mortality rate | 30 days
  Mortality rate
Duration on ICU | 30 days
  Duration on ICU measured in days
Reuptake on ICU | 30 days
  Reuptake on ICU and transferring ward
Handover duration patient | up to 3 months
  Handover duration per single patient
Handover duration entire | up to 3 months
  entire handover duration
Interruptions | up to 3 months
  Interruptions during handover categories: none, < 5min, > 5min
physicians satisfaction | through study completion, an average of 5 months
  evaluation of satisfaction by questionnaire
Change of SOFA Score at hour 72 | baseline and hour 72
  Change of SOFA Score to baseline (admission) and after 72 hours
Change of SOFA Score at hour 120 | baseline and hour 120
  Change of SOFA Score to baseline (admission) and after 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Marx, Prof., Study Chair — Uniklinik RWTH Aachen
Locations (1):
- RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] Keebler JR, Lazzara EH, Patzer BS, Palmer EM, Plummer JP, Smith DC, Lew V, Fouquet S, Chan YR, Riss R. Meta-Analyses of the Effects of Standardized Handoff Protocols on Patient, Provider, and Organizational Outcomes. Hum Factors. 2016 Dec;58(8):1187-1205. doi: 10.1177/0018720816672309. Epub 2016 Oct 17. PMID 27821676
- [Background] Starmer AJ, Landrigan CP; I-PASS Study Group. Changes in medical errors with a handoff program. N Engl J Med. 2015 Jan 29;372(5):490-1. doi: 10.1056/NEJMc1414788. No abstract available. PMID 25629753
- [Background] Starmer AJ, Spector ND, Srivastava R, West DC, Rosenbluth G, Allen AD, Noble EL, Tse LL, Dalal AK, Keohane CA, Lipsitz SR, Rothschild JM, Wien MF, Yoon CS, Zigmont KR, Wilson KM, O'Toole JK, Solan LG, Aylor M, Bismilla Z, Coffey M, Mahant S, Blankenburg RL, Destino LA, Everhart JL, Patel SJ, Bale JF Jr, Spackman JB, Stevenson AT, Calaman S, Cole FS, Balmer DF, Hepps JH, Lopreiato JO, Yu CE, Sectish TC, Landrigan CP; I-PASS Study Group. Changes in medical errors after implementation of a handoff program. N Engl J Med. 2014 Nov 6;371(19):1803-12. doi: 10.1056/NEJMsa1405556. PMID 25372088
- [Background] Starmer AJ, Sectish TC, Simon DW, Keohane C, McSweeney ME, Chung EY, Yoon CS, Lipsitz SR, Wassner AJ, Harper MB, Landrigan CP. Rates of medical errors and preventable adverse events among hospitalized children following implementation of a resident handoff bundle. JAMA. 2013 Dec 4;310(21):2262-70. doi: 10.1001/jama.2013.281961. PMID 24302089
- [Background] Randmaa M, Swenne CL, Martensson G, Hogberg H, Engstrom M. Implementing situation-background-assessment-recommendation in an anaesthetic clinic and subsequent information retention among receivers: A prospective interventional study of postoperative handovers. Eur J Anaesthesiol. 2016 Mar;33(3):172-8. doi: 10.1097/EJA.0000000000000335. PMID 26760400
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Kostoff M, Burkhardt C, Winter A, Shrader S. An Interprofessional Simulation Using the SBAR Communication Tool. Am J Pharm Educ. 2016 Nov 25;80(9):157. doi: 10.5688/ajpe809157. PMID 28090106
- [Background] Yee KC, Wong MC, Turner P. "HAND ME AN ISOBAR": a pilot study of an evidence-based approach to improving shift-to-shift clinical handover. Med J Aust. 2009 Jun 1;190(S11):S121-4. doi: 10.5694/j.1326-5377.2009.tb02617.x. PMID 19485859
- [Derived] Verholen N, Vogt L, Klasen M, Schmidt M, Beckers S, Marx G, Sopka S. Do Digital Handover Checklists Influence the Clinical Outcome Parameters of Intensive Care Unit Patients? A Randomized Controlled Pilot Study. Front Med (Lausanne). 2021 Apr 20;8:661343. doi: 10.3389/fmed.2021.661343. eCollection 2021. PMID 33959627
- See also: Patient Safety World Health Organisation — http://www.euro.who.int/en/health-topics/Health-systems/patient-safety
- See also: Data and Statistics Wold health Organisation — http://euro.who.int/en/health-topics/Health-systems/patient-safety/data-and-statistics
- See also: Australian Commission on Safety and Quality in Health Care — https://www.safetyandquality.gov.au/
- See also: Krankenhaus-Checkliste — https://www.weisse-liste.de/de/krankenhaus/checkliste/
- See also: Uniklinik RWTH Aachen — https://www.ukaachen.de